CLINICAL TRIAL: NCT00287872
Title: VELCADE (Bortezomib) and Thalidomide in Newly Diagnosed Patients With Multiple Myeloma
Brief Title: Bortezomib and Thalidomide in Treating Patients With Newly Diagnosed Stage II or Stage III Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0456 CDR0000450772; P30CA006973 (NIH); JHOC-J0456; JHOC-04063003; MILLENNIUM-JHOC-J0456
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2014-06

CONDITIONS: Multiple Myeloma
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib and Thalidomide (Experimental): The patients will receive Bortezomib on days 1, 4, 8 and 11 of each 21 day cycle in combination with daily oral Thalidomide.
  Interventions: Drug: bortezomib; Drug: thalidomide

INTERVENTIONS:
Drug: bortezomib
  Other Names: VELCADE
Drug: thalidomide

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Thalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. Giving bortezomib together with thalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with thalidomide works in treating patients with newly diagnosed stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor efficacy of bortezomib and thalidomide in patients with newly diagnosed stage II or III multiple myeloma.
* Determine the incidence and severity of peripheral motor/sensory neuropathy in patients treated with this regimen.
* Assess the ability to mobilize and collect stem cells in patients who undergo future autologous peripheral stem cell transplantation.
* Determine the time to response in patients treated with this regimen.
* Assess the quality of life of patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive bortezomib IV on days 1, 4, 8, and 11 and oral thalidomide once daily on days 1-21. Treatment repeats every 21 days for at least 4 courses. Patients who plan to undergo transplantation AND achieve ≥ 50% reduction in the tumor burden proceed to transplantation off study. Patients who do not undergo transplantation receive 2 additional courses of therapy beyond best response for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients who achieve at least a partial response after completion of treatment may receive maintenance therapy comprising bortezomib IV every 2 months and oral thalidomide* once daily OR twice every 2 months (i.e., the day before and the day of bortezomib administration) in the absence of disease progression or unacceptable toxicity.

NOTE: *For patients who had previously discontinued thalidomide, maintenance therapy may consist of bortezomib only.

Quality of life is assessed at baseline, at the beginning of each study course, and after completion of study treatment.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed Salmon-Durie stage II or III multiple myeloma

  * Untreated disease OR patient underwent prior therapy for this cancer that lasted no more than 2 weeks
* Measurable paraprotein in serum or urine (serum free-lite assay measurement allowed)
* No evidence of cord compression requiring concurrent steroids

PATIENT CHARACTERISTICS:

* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of contraception, including ≥ 1 highly effective method, 4 weeks before, during, and for ≥ 4 weeks after completion of study treatment
* No known HIV positivity
* No peripheral neuropathy ≥ grade 2
* No hypersensitivity to bortezomib, boron, or mannitol

PRIOR CONCURRENT THERAPY:

* No prior bortezomib
* More than 28 days since prior regimens with a duration of > 1 week but ≤ 2 weeks
* No steroids within 14 days prior to study entry
* No concurrent corticosteroids except for the treatment of a nonmalignant condition

  * May not exceed the equivalent dose of prednisone 10 mg/day
* No concurrent chemotherapy, immunotherapy, radiotherapy, or surgery
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borrello, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Ghosh N, Ye X, Ferguson A, Huff CA, Borrello I. Bortezomib and thalidomide, a steroid free regimen in newly diagnosed patients with multiple myeloma. Br J Haematol. 2011 Mar;152(5):593-9. doi: 10.1111/j.1365-2141.2010.08534.x. Epub 2011 Jan 17. PMID 21241279

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib and Thalidomide: The patients will receive Bortezomib on days 1, 4, 8 and 11 of each 21 day cycle in combination with daily oral Thalidomide.
  bortezomib
  thalidomide
Period: Overall Study
Arm/Group | Bortezomib and Thalidomide
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib and Thalidomide
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Treatment
Description: Clinical evaluations of disease response were determined with each cycle. Bone marrow biopsies were done at baseline and at study termination. Clinical responses were defined by the International Myeloma Working Group criteria: Stringent Complete Response (SCR), CR and normal free light chain ratio and no clonal cells in bone marrow; Complete Response (CR), Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; Very Good Partial Response (VGPR), Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; Partial Response (PR), ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. Objective response is defined as a best overall response of SCR, CR, VGPR, or PR.
Time Frame: 1-6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib and Thalidomide
Number analyzed (Participants) | 27
percentage of participants | 81.5 [62 to 94]

2. Secondary Outcome: Peripheral Motor and Sensory Neuropathy (Grade 2 and Higher)
Description: Neuropathy was monitored using Total Neuropathy Score reduced (TNSr).
Time Frame: 1-6 months
Measure: Number; unit: participants
Arm/Group | Bortezomib and Thalidomide
Number analyzed (Participants) | 27
participants | 19

3. Secondary Outcome: Mobilization of Stem Cells in Patients Proceeding to Autologous Peripheral Stem Transplantation
Time Frame: 1-6 months
Population: Analysis not completed as the information was not relevant since no patients went on to transplant.
Arm/Group | Bortezomib and Thalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: The Time to Response
Time Frame: 1-6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib and Thalidomide
Number analyzed (Participants) | 22
months | 2 [0.5 to 5.8]

5. Secondary Outcome: Quality of Life
Time Frame: 0-6 months
Population: Analysis not done on subject population.
Arm/Group | Bortezomib and Thalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Bortezomib and Thalidomide
Serious Adverse Events (participants affected / at risk) | 10/30
Other Adverse Events (participants affected / at risk) | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Thalidomide (N=30)
dehydration (Gastrointestinal disorders) | 2 (2)
nausea & vomiting (Gastrointestinal disorders) | 2 (2)
renal failure (Renal and urinary disorders) | 1 (1)
neutropenic fever (Infections and infestations) | 1 (1)
pneumonia (Infections and infestations) | 3 (3)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Thalidomide (N=30)
peripheral neuropathy (Nervous system disorders) | 25 (75)
hypotension (Cardiac disorders) | 6 (7)
fatigue (General disorders) | 22 (48)
constipation (Gastrointestinal disorders) | 19 (40)
diarrhoea (Gastrointestinal disorders) | 15 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes